CLINICAL TRIAL: NCT05302479
Title: Validating the Modified COMPASS 31 Questionnaire for Evaluation and Outcomes of Post-concussive Symptoms in Active Duty Military Patients
Brief Title: Validating a Modified COMPASS 31questionnaire for Treatment Outcomes
Acronym: COMPASS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: The Defense and Veterans Brain Injury Center (U.S. Federal Agency); The University of Queensland (Other)
Responsible Party: Principal Investigator, Matt Hammerle, Doctor of Physical Therapy, Brooke Army Medical Center
Other Study IDs: C.2021.128e
Record Dates: First submitted 2022-02-23; First posted 2022-03-31 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Headache, Migraine; Persistent Post Traumatic Headache; Cervicogenic Headache
MeSH Terms: conditions — Migraine Disorders; Post-Traumatic Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: COMPASS 31 questionnaire — A 31 question questionnaire that measures autonomic symptoms.

SUMMARY:
Eligible participants will complete the COMPASS 31 (year), modified COMPASS 31(one month) and the NSI (one month) questionnaires at baseline and complete the modified COMPASS 31 and the NSI after usual care of treatment.

The investigators will

1. Compare results for the COMPASS 31(year) to the modified COMPASS 31(month) at baseline.
2. Compare modified COMPASS 31(month) to the NSI at baseline and post intervention.

DETAILED DESCRIPTION:
The Composite Autonomic Symptom Score (COMPASS 31) is a validated questionnaire designed to measure self reported autonomic symptoms in the last year in individuals with migraine and post-concussive symptoms. In order to use this questionnaire to measure response to treatment it would be preferable to determine if the results of the COMPASS 31 are similar if the patient is asked to complete this thinking about symptoms in the last year as per the usual questionnaire, compared to a modified COMPASS 31 where symptoms in the past month will be assessed.

This prospective trial will compare results of the COMPASS 31 (year) to the modified COMPASS 31 (month). Since the present gold standard for outcome measures in post-concussive treatment is the neurobehavioral symptom inventory (NSI), this study will also compare results of the modified COMPASS 31(month) to the NSI outcome measure at baseline and post treatment to validate the utilization of the modified version of the COMPASS 31(month) for use in the post-concussive population as an outcome measure for self-reported autonomic nervous system symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the BAMC_BIRS clinic for treatment of headache between the ages of 18-64.

Exclusion Criteria:

* Normal composite autonomic symptom score.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who present for treatment of headache in the military medical clinic tend to be active duty military patients however retirees and family members will not be excluded from participation.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Composite Autonomic Symptom Score questionnaire (Compass 31)-Self reported autonomic nervous system symptoms in the past year. | One year
  Self reported autonomic nervous system symptoms in the past year will be measured using the validated, refined and abbreviated Composite Autonomic Symptom Score questionnaire (Compass 31). Scoring ranges from 0-100 with higher scores indicating more autonomic symptoms.
Composite Autonomic Symptom Score questionnaire (Compass 31)- Self reported autonomic nervous system symptoms in the past month (COMPASS 31-month). | One month
  Self reported autonomic nervous system symptoms in the past month will be measured using the validated, refined and abbreviated Composite Autonomic Symptom Score questionnaire (Compass 31-month). Scoring ranges from 0-100 with higher scores indicating more autonomic symptoms.
Neurobehavioural symptom inventory (NSI) a 22-item self-report questionnaire of neurobehavioral symptoms. | One month
  Neurobehavioural symptom inventory (NSI) a 22-item self-report questionnaire of neurobehavioral symptoms. Scores range from 0-88 with higher scores indicating more symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Matt H Hammerle, DPT, Principal Investigator — BAMC-BIRS
Locations (1):
- Brooke Army Medical Centre, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howard L, Dumkrieger G, Chong CD, Ross K, Berisha V, Schwedt TJ. Symptoms of Autonomic Dysfunction Among Those With Persistent Posttraumatic Headache Attributed to Mild Traumatic Brain Injury: A Comparison to Migraine and Healthy Controls. Headache. 2018 Oct;58(9):1397-1407. doi: 10.1111/head.13396. Epub 2018 Aug 29. PMID 30156267
- [Background] King PR, Donnelly KT, Donnelly JP, Dunnam M, Warner G, Kittleson CJ, Bradshaw CB, Alt M, Meier ST. Psychometric study of the Neurobehavioral Symptom Inventory. J Rehabil Res Dev. 2012;49(6):879-88. doi: 10.1682/jrrd.2011.03.0051. PMID 23299259